CLINICAL TRIAL: NCT01532986
Title: Improving Quality of Care in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Randomized Trial to Test the "Coordinated Care for Health Promotion and Activities in Parkinson's Disease" Intervention in the VA
Acronym: CHAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRI 11-126
Record Dates: First submitted 2012-01-13; First posted 2012-02-15 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease
Keywords: Quality of Health Care; Nursing Care Management; Care Coordination; Randomized Trials
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Arm 1) (Other): Veterans randomized to the usual care arm will continue to receive care they would have received if they had not enrolled in the study; no care or resources that are made available in general by VA will be withheld from participants in either arm or to any Veterans who wish to use those resources.
  Educational handout: brief educational handout on Parkinson's disease that is available in the VA's "Healthwise for Life" handbook.
  Interventions: Other: Coordinated care management for Parkinson's disease; Other: Educational handout
- Intervention (Arm 2) (Experimental): A delivery system redesign, with nurse care managers, using standardized assessment tools and care coordination protocols to address unmet needs of Veterans with Parkinson's Disease (PD) by collaborating with these Veterans and their families, providers, and community partners.
  Educational handout: brief educational handout on Parkinson's disease that is available in the VA's "Healthwise for Life" handbook.
  Interventions: Other: Coordinated care management for Parkinson's disease

INTERVENTIONS:
Other: Coordinated care management for Parkinson's disease — Nurse care managers will use standardized assessment tools and care coordination protocols to address unmet needs of Veterans with PD, and collaborate with these Veterans and their families, providers, and community partners to manage PD care.
Other: Educational handout — To minimize potential bias from participants' awareness of randomization arm assignment, the investigators will provide to all study participants (intervention arm and usual care arm) on enrollment a brief educational handout on Parkinson's disease that is available in the VA's "Healthwise for Life" handbook (page 273). This information includes a definition of PD, its symptoms, and several suggestions for managing PD such as medications and regular exercise.
  Arms: Usual Care (Arm 1)

SUMMARY:
Health care benefits and services are received through the Veterans Health Administration (VHA), a component of the United States Department of Veterans Affairs. Over 40,000 Veterans across the Veterans Health Administration are diagnosed with Parkinson's disease (PD), a chronic condition that affects motor function as well as cognition, mood, sleep, and autonomic function. There are not enough subspecialists to manage every Veteran with Parkinson's disease. However, a care model of nurse care managers as catalysts and advocates using needs assessments, evidence-based protocols, and VHA and community access coordination mechanisms to optimize Parkinson's disease care may improve quality of Parkinson's disease care and patient-centered outcomes. If efficacious, this model may be practical to disseminate via an existing VHA national consortium network for Parkinson's disease.

Objectives are (1) to implement then analyze via a randomized controlled trial whether a nurse-led, coordinated care management intervention, Care Coordination for Health Promotion and Activities in Parkinson's Disease (CHAPS), compared to usual care will improve adherence to evidence-based practice guidelines and improve health outcomes in Veterans with Parkinson's disease in a region of the southwest United States, and (2) to analyze extent of implementation of the CHAPS intervention and its costs to determine how the intervention can be made sustainable and disseminated throughout Veterans Affairs Medical Centers if efficacious.

DETAILED DESCRIPTION:
In a 5-year randomized controlled trial, we enrolled 345 Veterans with PD that were then randomized in a 1:1 ratio to receive up to 24 months of a PD care management program, "Care Coordination for Health Promotion and Activities in Parkinson's Disease" (CHAPS), or continue with usual care. Eligible participants across 5 sites of the Southwest Parkinson's Disease Research, Education and Clinical Center (SW PADRECC): Greater Los Angeles, Las Vegas, Loma Linda, Long Beach and San Diego VISN 22 (VA Desert Pacific Healthcare Network) facilities were identified through administrative data and vetted by physicians. The multi-faceted nurse-led intervention, CHAPS, incorporated PD quality improvement (QI) tools to enhance proactive Veteran-centered care delivery. PDQI tools included: (1) a structured telephone assessment administered by a nurse care manager (NCM) to proactively identify medical problems and unmet needs; (2) problem-specific evidence-based interventions organized into treatment plans including follow-up/monitoring protocols with VA and community linkages; (3) the Siebens Domain Management ModelTM, a structural approach to improve collection and organization of health information and enrich communication among providers; (4) Siebens Health Care Notebooks prepared with Veteran self-management materials; (5) a Microsoft Access care management database, containing the CHAPS Assessment and algorithms for problem identification based on Veteran data; and (6) decision-support meetings of NCMs with movement disorder specialists. Research interviewers administer a structured telephone survey at baseline, 6, 12, 18, and 24 months. Participants were provided $25 per survey. Medical records were abstracted.

Ongoing analyses (1) measure PD quality indicator adherence, health outcomes, and health service utilization; (2) evaluate qualitative and quantitative data to summarize the extent of intervention implementation and barriers and facilitators to potential dissemination; and (3) examine costs of CHAPS care and cost offset between randomization arms to provide new knowledge to aid in future dissemination of the CHAPS Program in a "National Rollout" according to the VA Quality Enhancement Research Initiative QUERI process.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the United States of America
* Receiving health care at one of five Veterans Health Administration medical centers in the southwest United States: Greater Los Angeles, Loma Linda, Long Beach, or San Diego, California, or Las Vegas, Nevada.
* Diagnosis of Parkinson's disease (PD)
* At least two ICD-9 diagnostic codes for PD (332.0) in the administrative data from October 1, 2010 - to present date or until recruitment target is met
* At least 18 years of age
* Must demonstrate capacity to provide consent for study participation.

Exclusion Criteria:

* Any Veteran who is a study subject in the Deep Brain Stimulation (DBS) VA cooperative study as these subjects are not to enroll in any other study per DBS study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Connor, PhD RN MBA, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (5):
- United States (5):
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Connor K, Cheng E, Siebens HC, Lee ML, Mittman BS, Ganz DA, Vickrey B. Study protocol of "CHAPS": a randomized controlled trial protocol of Care Coordination for Health Promotion and Activities in Parkinson's Disease to improve the quality of care for individuals with Parkinson's disease. BMC Neurol. 2015 Dec 15;15:258. doi: 10.1186/s12883-015-0506-y. PMID 26670300
- [Derived] Connor KI, Siebens HC, Mittman BS, Ganz DA, Barry F, McNeese-Smith DK, Cheng EM, Vickrey BG. Implementation fidelity of a nurse-led RCT-tested complex intervention, care coordination for health promotion and activities in Parkinson's disease (CHAPS) in meeting challenges in care management. BMC Neurol. 2022 Jan 24;22(1):36. doi: 10.1186/s12883-021-02481-5. PMID 35073865
- [Derived] Connor KI, Siebens HC, Mittman BS, McNeese-Smith DK, Ganz DA, Barry F, Edwards LK, McGowan MG, Cheng EM, Vickrey BG. Stakeholder perceptions of components of a Parkinson disease care management intervention, care coordination for health promotion and activities in Parkinson's disease (CHAPS). BMC Neurol. 2020 Dec 2;20(1):437. doi: 10.1186/s12883-020-02011-9. PMID 33267827
- [Derived] Connor KI, Siebens HC, Mittman BS, Ganz DA, Barry F, Ernst EJ, Edwards LK, McGowan MG, McNeese-Smith DK, Cheng EM, Vickrey BG. Quality and extent of implementation of a nurse-led care management intervention: care coordination for health promotion and activities in Parkinson's disease (CHAPS). BMC Health Serv Res. 2020 Aug 10;20(1):732. doi: 10.1186/s12913-020-05594-8. PMID 32778083
- [Derived] Connor KI, Cheng EM, Barry F, Siebens HC, Lee ML, Ganz DA, Mittman BS, Connor MK, Edwards LK, McGowan MG, Vickrey BG. Randomized trial of care management to improve Parkinson disease care quality. Neurology. 2019 Apr 16;92(16):e1831-e1842. doi: 10.1212/WNL.0000000000007324. Epub 2019 Mar 22. PMID 30902908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 345 participants enrolled in the study. Subjects were identified by a treating provider while receiving care at 5 Veterans Administration health systems.
Pre-assignment Details: 13 removed before baseline survey. 4 were ineligible due to not having Parkinson's disease. This left 328 who were randomized
Period: Overall Study
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Started | 166 | 162
Completed | 143 | 138
Not Completed | 23 | 24
Not completed — Death | 9 | 9
Not completed — Withdrawal by Subject | 7 | 10
Not completed — Physician Decision | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Usual Care (Arm 1); Intervention (Arm 2): A delivery system redesign, with nurse care managers, using standardized assessment tools and care coordination protocols to address unmet needs of Veterans with Parkinson's Disease (PD) by collaborating with these Veterans and their families, providers, and community partners.
  Educational handout: brief educational handout on Parkinson's disease that is available in the VA's "Healthwise for Life" handbook.
- Total: Total of all reporting groups
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2) | Total
Number analyzed (Participants) | 166 | 162 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.2) | 69.6 (10.1) | 70.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 164 | 155 | 319
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American/Black | 11 | 9 | 20
  Asian-American | 0 | 3 | 3
  American-Indian/Alaskan Native | 3 | 2 | 5
  Caucasian/White | 131 | 125 | 256
  Hispanic/Latino | 16 | 21 | 37
  Native Hawaiian/Other Pacific Islander | 3 | 0 | 3
  More than One Race | 1 | 0 | 1
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Measures Adhered To in the PD Guidelines
Description: Adherence to quality measures for Parkinson's disease care during study period. We operationalized 18 quality measures: 12 were determined through chart review, and 6 were measured using patient survey data.
  Range and direction of score: 0 (worst) to 1 (best)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: proportion of quality measures followed
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
proportion of quality measures followed | 0.77 (0.16) | 0.58 (0.14)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.189, 95% CI 2-sided [0.157 to 0.222]

2. Secondary Outcome: Health Utilities Index (HUI3)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: -0.36 (worst) to 1 (best)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 0.48 (0.3) | 0.43 (0.3)
  6 months | 0.46 (0.3) | 0.44 (0.3)
  12 months | 0.44 (0.3) | 0.42 (0.3)
  18 months (final) | 0.40 (0.3) | 0.40 (0.3)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.04 to 0.08]

3. Secondary Outcome: Activities of Daily Living (ADL), (Speech and Swallowing Only)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: 0 (best) to 16 (worst)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 4.44 (2.9) | 4.68 (3.1)
  6 months | 4.48 (3.0) | 4.75 (3.1)
  12 months | 4.96 (3.2) | 5.06 (3.1)
  18 months (final) | 5.02 (3.3) | 5.35 (3.2)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.52 to 0.57]

4. Secondary Outcome: Medical Outcomes Study (MOS)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: 1 (worst) to 5 (best)
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 3.91 (0.9) | 4.07 (0.8)
  6 months | 3.93 (0.9) | 3.91 (0.8)
  12 months | 3.91 (0.9) | 4.00 (0.8)
  18 months (final) | 3.94 (0.9) | 4.03 (0.7)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.34 to 0.10]

5. Secondary Outcome: General Self-Efficacy Scale (GSES)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: 10 (worst) to 40 (best)
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 33.97 (5.1) | 34.17 (5.5)
  6 months | 34.74 (4.9) | 34.34 (5.6)
  12 months | 35.07 (5.1) | 34.38 (5.7)
  18 months (final) | 35.1 (5.1) | 34.04 (5.9)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-2.04 to 0.29]

6. Secondary Outcome: Consumer Assessment of Healthcare Providers and Systems (CAHPS)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: 0 (worst) to 100 (best)
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 58.72 (33.4) | 53.42 (34.9)
  6 months | 60.18 (32.6) | 55.34 (33.6)
  12 months | 58.25 (34.2) | 54.16 (34.5)
  18 months (final) | 58.55 (33.6) | 53.66 (35.0)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.22, 95% CI 2-sided [-8.02 to 10.46]

7. Secondary Outcome: Patient Assessement of Care for Chronic Conditions (PACIC)
Description: as for outcome 4
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baselin | 2.34 (0.9) | 2.15 (0.8)
  6 months | 2.28 (0.8) | 2.16 (0.7)
  12 months | 2.32 (0.8) | 2.28 (0.8)
  18 months (final) | 2.37 (0.8) | 2.30 (0.8)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.00 to 0.34]

8. Secondary Outcome: World Health Organization Well-Being Index (WHO-5)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Range and direction of score: 1 (worst) to 25 (best)
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
units on a scale
  Baseline | 14.19 (5.8) | 13.14 (5.9)
  6 months | 15.02 (5.7) | 13.93 (5.9)
  12 months | 14.20 (6.0) | 13.38 (6.5)
  18 months (final) | 14.14 (6.3) | 13.45 (6.5)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.45 to 1.33]

9. Secondary Outcome: Percentage With a Patient Healthcare Questionnaire-2 (PHQ-2) Score ≥ 3
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  PHQ-2 score ranges from 0 to 4. Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  Higher scores indicate detection of depressive symptoms
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 166 | 162
Participants
  Baseline | 13 | 22
  6 months | 15 | 13
  12 months | 11 | 16
  18 months (final) | 23 | 11
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -11.52, 95% CI 2-sided [-20.42 to -2.62]

10. Secondary Outcome: Patient Healthcare Questionnaire-9 (PHQ-9)
Description: Data collected at baseline, 6, 12, 18 months. Missing values imputed by last-value carried forward.
  Range and direction of score: 0 (best) to 27 (worst). Reported results compared compared data of baseline and final survey results. Additional analyses included repeated-measures models that included data from all time points.
  PHQ-9 was only administered to subjects who had a score of 3 or higher on the PHQ-2
Time Frame: 18 months
Population: PHQ-9 was only administered to subjects who had a score of 3 or higher on the PHQ-2. At baseline, this was only 13 persons in usual care and 22 persons in the intervention group
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
Number analyzed (Participants) | 13 | 22
units on a scale
  Baseline | 12.33 (4.4) | 14.45 (3.9)
  6 months | 12.96 (4.8) | 13.22 (4.2)
  12 months | 12.44 (4.2) | 12.97 (3.6)
  18 months (final) | 12.21 (4.8) | 12.46 (4.1)
Statistical Analysis 1: Comparison: Usual Care (Arm 1) vs Intervention (Arm 2); Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-4.20 to 0.24]

ADVERSE EVENTS:
Time Frame: 18 months
Description: Because this is a care intervention to promote best practices, we do not believe that deaths observed to this study should be considered adverse events of the study.
Arm/Group | Usual Care (Arm 1) | Intervention (Arm 2)
All-Cause Mortality (participants affected / at risk) | 9/166 | 9/162
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/162
Other Adverse Events (participants affected / at risk) | 0/166 | 0/162

LIMITATIONS AND CAVEATS:
Study implemented within the Veterans Administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT01532986/Prot_SAP_000.pdf